CLINICAL TRIAL: NCT04341246
Title: Characterization and Technical Evaluation of cT1 for NASH (CATE-NASH): A Case-control Study
Brief Title: Characterization and Technical Evaluation of cT1 for NASH (CATE-NASH)
Status: Completed | Type: Observational
Sponsor: Perspectum (Industry)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: IIP-174
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: NASH; Livermultiscan; fatty liver
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Cases: Cases are defined as those patients who have undergone liver biopsy and have confirmed NASH and fibrosis
  Interventions: Device: LiverMultiscan
- Controls: Controls are patients have undergone a liver biopsy with neither significant NASH nor significant fibrosis
  Interventions: Device: LiverMultiscan

INTERVENTIONS:
Device: LiverMultiscan — The Livermultiscan is a quick, 15 minute contrast free MRI scan that provided metrics to quantify liver health namely fat, iron and fibro-inflammation
  Other Names: LMS

SUMMARY:
The primary objective of this study is to evaluate to provide evidence to establish tightly defined cut-offs to identify patients for NASH clinical trial inclusion using cT1 and/or PDFF. The study will be divided into 2 sub groups comprising of cases and controls.

DETAILED DESCRIPTION:
This is a prospective, case-control, study designed to measure the mean difference in cT1 and PDFF in patients who have undergone liver biopsy and have confirmed NASH and fibrosis or 'cases' (N=40) and N=20 patients with neither significant NASH nor significant fibrosis 'controls'.

Confirmed cases will be patients who have met the criteria for active NASH with fibrosis according to the NAS CRN scoring system (NAS≥4 & F2-3), 'controls' will be those who did not meet NASH diagnostic criteria and have evidence of fibrosis of ≤2.

In addition, in order to investigate the variability of the biomarker investigators will assess the 'measurement' error in all participants by performing a repeat 'second' scan in the same scanning session, and , in cases only, 'biological' variability by performing a repeat scan in controls 2-4 weeks later.

Suitable patients based on trial inclusion criteria will be identified by the study PI and clinical collaborator and invited to receive one or two MRI scans from which cT1 and PDFF will be derived using Perspectum's LiverMultiScan software. Baseline scan will ideally be performed between 3 days (to allow for recovery from the procedure and time for biopsy results to become available) and 6 weeks following biopsy, to minimize the likelihood that the patient is in a significantly different pathophysiologic state on the baseline scan day than on the biopsy day.

In order to ensure that the investigators capture information on normal variability and not related to intervention they will also capture and record basic information at both measurement timepoints (e.g. body weight, waist circumference, details of lifestyle interventions).

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged between 18-75 years
* Ability to understand and sign a written informed consent form (ICF)
* Patients who have undergone a liver biopsy within the last 6 weeks because of clinical suspicion on NAFL-D

Exclusion Criteria:

* Prior or planned liver transplantation
* Patients who have undergone a laparoscopic or wedge liver biopsy, or biopsy taken from the left lobe
* Participation in an investigational new drug (IND) trial in the 30 days before enrolment (except those patients who were not administered the IND)
* Other known causes of chronic liver disease based on clinical criteria at the study site, such as the following:

  * Alcoholic liver disease
  * Primary biliary cirrhosis
  * Primary sclerosing cholangitis
  * Autoimmune hepatitis
  * Wilson's disease, hemochromatosis, iron overload
  * Alpha-1-antitrypsin (A1AT) deficiency
  * Hepatitis C Virus, Hepatitis B Virus
* History or diagnosis of cirrhosis and/or hepatic decompensation including ascites, hepatic encephalopathy or variceal bleeding
* Clinically relevant (more than 3 drinks per day on average for men and 2 for women) alcohol abuse within 12 months of liver biopsy and/or any recreational drugs
* Any contradiction or significant limitation to Magnetic Resonance imaging (MRI) scanning including but not limited to the following:

  * Claustrophobia preventing Magnetic Resonance imaging (requires 15-30 minutes in scanner)
  * Pacemaker or another implanted electronic device
  * Metal in body (such as aneurysm clip) that might produce artefact on abdominal MRI or might be adversely impacted by a high magnetic field
  * Inability to lie flat, remain till, or briefly hold breath as necessary during MR imaging
  * Medical condition likely to produce significant hypervolemia like congestive heart failure
  * Severe obesity complicating positioning within MR scanner
* Concomitant medical illnesses per investigators discretion that would hamper patient's completion of the study or otherwise affect the collected data (such as HIV infection, recent major surgery, uncontrolled heart disease, concurrent infection or fever of unknown origin, illicit drug use, cancer)
* Clinically significant medical or psychiatric condition considered a high risk for participation in an investigational study
* Failure to give informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, deemed to be suitable for inclusion into a NASH clinical trial based on their clinical risk factors, and who have been referred for a standard of care diagnostic liver biopsy on suspicion of NASH
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-12 (Actual)

PRIMARY OUTCOMES:
To demonstrate that a binary decision algorithm applied to cT1 can significantly identify patients whose liver biopsy results would qualify them for randomization in a clinical trial testing an investigational treatment for NASH | 6 weeks
  Mean cT1 (and PDFF) values for those with NAS≥4&F2-3 (cases) and those with NAS<4 or F<2 (controls)

SECONDARY OUTCOMES:
To determine the measurement test-retest repeatability of cT1 and PDFF in the target patient population by examining the test-retest variability within a single scanning session | 1 day
  Difference between two replicates (Scan A and Scan B in same session) under the same measurement conditions expressed as the repeatability coefficient
To determine the biological repeatability of cT1 and PDFF in the target patient population by examining the test-retest variability between scans acquired under the same conditions but 2-4 weeks apart | 2-4 weeks
  Difference between two scans (Scan 1 and Scan 2) under the same measurement conditions expressed as the repeatability coefficient

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen, Corey,, MD, MPH, MMSc, Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided